CLINICAL TRIAL: NCT07267520
Title: The Effects of Quartz Crystal Singing Bowl Music and Guided Relaxation on Mood and Sleep in Young Adults
Brief Title: The Effects of Quartz Crystal Singing Bowl Music and Guided Relaxation on Mood and Sleep in Rangatahi (Young Adults)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Waikato (Other)
Collaborators: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Nicola Starkey, Professor of Psychology, The University of Waikato
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HREC(Health)2024#3
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy Young Adults
Keywords: Mood; Crystal singing bowls; Progressive muscle relaxation; online intervention
MeSH Terms: interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quartz Crystal Singing Bowls music (Experimental)
  Interventions: Behavioral: Quartz Crystal Singing Bowl music
- Progressive Muscle Relaxation (Active Comparator)
  Interventions: Behavioral: Progressive Muscle Relaxation

INTERVENTIONS:
Behavioral: Quartz Crystal Singing Bowl music — The quartz crystal singing bowls audio track used in the current study was "Tranquility" by Annie Jameson. The audio track was 570 seconds (9.5 minutes) for all sessions. Annie Jameson composed the track herself and gave permission for its use. The full Tranquility track can be found on YouTube (https://www.youtube.com/watch?v=0mX3Vqvo5k4) or Spotify. The audio was accessed online via the Qualtrics platform
  Arms: Quartz Crystal Singing Bowls music
Behavioral: Progressive Muscle Relaxation — A guided progressive muscle relaxation audio (recorded by the NZ Cancer Society https://www.youtube.com/watch?v=Zydrp3rfJdY) and similar to the PMR script from the Anxiety and Phobia Workbook by Edmund Bourne was used. The session took approximately 12 minutes. Participants were instructed to start by sitting or lying comfortably, taking some deep breaths and then tense and relax muscles in a sequential manner from the head to the feet. The audio was presented online via Qualtrics software
  Arms: Progressive Muscle Relaxation

SUMMARY:
The number of people reporting poor mental wellbeing is increasing, with rates exceeding 25% of the population. Rates of psychological distress in young people (aged 15-24 years) are rapidly increasing but many cannot access professional help. Self-help options such as meditation and mindfulness are effective in decreasing stress and enhancing mood, but time, practice, self-motivation and patience are required to fully realise the benefits. Thus, there is a need to explore alternate treatment options.

This study seeks to determine if the effects of listening to quartz crystal singing bowl music (CSBs) are equivalent to that of progressive guided muscle relaxation on self-report measures of mood, stress and sleep in young adults at 4- and 8- weeks post intervention. The intervention will be delivered online.

The main question it aims to answer is:

Are the effects of listening to singing bowl music equivalent to that of progressive guided muscle relaxation (PMR) on self-report measures of mood in young adults (Total Mood Disturbance of the POMS) at 4- and 8- weeks post intervention.

Does listening to singing bowls result in improved sleep and stress, similar to the effects of PMR.

Participants will be allocated to either the singing bowls or progressive muscle relaxation group. They will be sent a link to listen to the intervention 3 times a week for the first 4 weeks, and then weekly for the next 4 weeks. They will be asked to compete an online questionnaire at baseline, 4 weeks and 8 weeks.

At the end of the trial (8 weeks), participants will be given access to both singing bowls and progressive muscle relaxation interventions to use as often as they like.

ELIGIBILITY:
Inclusion Criteria:

* age 16-25 years

Exclusion Criteria:

* undergoing psychiatric/psychological treatment
* participation in guided relaxation more than once a month
* listened to singing bowls more than once a month

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 108 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in total mood disturbance (TMD) score between baseline, 4 weeks and 8 weeks | Baseline, 4 weeks and 8 weeks
  The TMD is derived from the profile of mood states questionnaire (abbreviated version). Participants are presented with a list of 40 words that describe feelings people have. They are asked to circle the number that best describes how they feel right now from 0 (not at all), 1 (a little), 2 (moderately), 3 (quite a lot) to 4 (extremely). Seven subscales are calculated by summing the relevant items (Tension, Anger, ERA-score range 0-24; Fatigue, Vigour, Confusion- score range 0-20; Depression - score range 0-28 ). A Total Mood Disturbance score (TMD) is also calculated by summing the totals for the negative subscales (Tension, Depression, Anger, Fatigue, Confusion), and subtracting the totals for the positive scales (Vigour, Esteem-related Affect). A constant (100) can be added to eliminate negative values. Scores (including the constant) range from 52-216. A higher score reflects a more negative mood state
Change in total mood disturbance (TMD) score between baseline, 4 weeks and 8 weeks | Baseline, 4 weeks and 8 weeks
  The TMD is derived from the profile of mood states questionnaire (abbreviated version). Participants are presented with a list of 40 words that describe feelings people have. They are asked to circle the number that best describes how they feel right now from 0 (not at all), 1 (a little), 2 (moderately), 3 (quite a lot) to 4 (extremely). Seven subscales are calculated by summing the relevant items (Tension, Anger, Fatigue, Depression, Esteem related affect, Vigour and Confusion). A Total Mood Disturbance score (TMD) is also calculated by summing the totals for the negative subscales (Tension, Depression, Anger, Fatigue, Confusion), and subtracting the totals for the positive scales (Vigour, Esteem-related Affect [Note that 2 items are reverse scored for the ERA subscale]. A higher score reflects a more negative mood state

SECONDARY OUTCOMES:
Change in POMS subscale scores at 4 and 8 weeks | Baseline, 4 weeks and 8 weeks
  The POMS has seven subscales: Tension, Anger, Fatigue, Depression, Esteem related affect, Vigour and Confusion. For the negative subscales (Tension, fatigue, confusion, depression and anger), a higher score indicates poorer mood. For the positive subscales (vigour and esteem related affect), a high score indicates a more positive mood.
Overall sleep quality | Baseline, 4 weeks, 8 weeks
  Rating of overall sleep quality from the Auckland Sleep questionnaire. Higher ratings (on a 1-4 scale) indicate poorer sleep quality
Visual analogues scales - immediately before and after a session | Once a week for 8 weeks
  To assess the acute effects of the intervention, participants will be asked to complete ratings of overall mood, relaxation, and stress before and after one session one session each week. Participants are asked to rate how they are feeling right now using a visual analogue scale (VAS) from 0 (worst I've ever felt not relaxed, not stressed,) to 100 (very stressed, very relaxed, best I've ever felt)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola J Starkey, Starkey, Principal Investigator — University of Waikato; Michael Jameson, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- School of Psychological and Social Sciences, Hamilton, Waikato Region, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
All data are available from the PI upon reasonable request
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months after publication with no end date
Access Criteria: Data can be obtained by emailing the PI with a proposal for planned analyses. The request will be reviewed by the co-PIs.

REFERENCES:
- [Background] Goldsby TL, Goldsby ME, McWalters M, Mills PJ. Effects of Singing Bowl Sound Meditation on Mood, Tension, and Well-being: An Observational Study. J Evid Based Complementary Altern Med. 2017 Jul;22(3):401-406. doi: 10.1177/2156587216668109. Epub 2016 Sep 30. PMID 27694559
- [Background] Matthews A, Phillips MC, Matthews LR, Kumar S, Pillai A, Jameson MB. A Pilot Study Evaluating the Effects of Relaxation Music Played on Quartz Crystal Singing Bowls on Mood in Teenage Males. J Psychiatry Behav Sci. 2023;6(2):1085

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-04-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT07267520/Prot_SAP_ICF_000.pdf